CLINICAL TRIAL: NCT03891329
Title: BIO|MASTER.Cor Family Study
Brief Title: Master Study of the Acticor/Rivacor ICDs/CRT-Ds and the Plexa ProMRI S DX Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TA115
Record Dates: First submitted 2019-02-11; First posted 2019-03-27 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Tachyarrhythmia
MeSH Terms: conditions — Heart Failure; Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acticor/Rivacor ICDs/CRT-Ds (Other): Implant of the new Cor Family internal cardioverter defibrillators (ICDs) / Cardiac Resynchronisation Therapy-Defibrillators (CRT-Ds) and Plexa ProMRI S DX lead (if applicable). Device measurements, pre-defined programming and Adverse Event Reporting
  Interventions: Device: Acticor/Rivacor ICDs/CRT-Ds; Device: Plexa S DX

INTERVENTIONS:
Device: Acticor/Rivacor ICDs/CRT-Ds — pre-defined device programming, measurements and follow-up schedule
Device: Plexa S DX — Implantation, measurements and follow-up schedule

SUMMARY:
Post-Market Clinical Follow-up of the new Cor Family ICDs/CRT-Ds (Acticor, Rivacor) and the new Plexa ProMRI S DX right ventricular lead to provide post-market data and supporting evidence for the clinical safety and performance of the devices.

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for ICD or CRT-D therapy according to clinical guidelines
* Planned for de novo implantation of an ICD/CRT-D, or upgrade/exchange from existing ICD/CRT-D or pacemaker implant
* Able to understand the nature of study and to provide written informed consent
* Willing and able to perform all follow-up visits at the study site
* Willing and able to use the CardioMessenger and accepts the BIOTRONIK Home Monitoring concept

Exclusion Criteria:

* Contraindication to ICD and CRT-D therapy
* Planned for implantation of a CRT-DX system
* For VR-T DX devices: permanent atrial tachyarrhythmia
* For VR-T DX devices: patients requiring atrial pacing
* Less than 18 years old
* Pregnant or breast feeding
* Participating in another interventional clinical investigation
* Life-expectancy is less than 12 months
* Cardiac surgical procedure planned within 12 months after implantation (including interventional procedures like ablation, valve replacement, heart transplant etc.). Procedures to occur during or prior to implantation are not exclusionary

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Steffel, MD, Principal Investigator — Universitätsspital Zürich
Locations (13):
- Kepler Universitätsklinikum, Linz, Austria
- Germany (4):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Charité Universitätsmedizin Berlin, Berlin
  - SRH Wald-Klinikum Gera GmbH, Gera
  - SRH Zentralklinikum Suhl, Suhl
- Hungary (2):
  - National Hospital of Cardiology, Balatonfüred
  - Semmelweis Medical University, Budapest
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Netherlands (2):
  - Hospital Medisch Spectrum Twente, Enschede
  - Erasmus Medical Center, Rotterdam
- East-Slovak Cardiology Institute (VUSCH), Košice, Slovakia
- Switzerland (2):
  - Inselspital - Universitätsspital Bern, Bern
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 130 patients completed the informed consent process and signed the informed consent sheet.
Pre-assignment Details: 127 patients received one or more study devices implanted. 3 enrolled patients did not receive a study device. Two of those patients who did not receive a study were excluded from the analysis while the third patient underwent an implantation attempt and was therefore included in the general analysis population
Groups:
- Acticor/Rivacor ICDs/CRT-Ds: Implant of the new Cor Family ICDs and Plexa ProMRI S DX lead (if applicable). Device measurements, pre-defined programming and Adverse Event Reporting
  Acticor/Rivacor ICDs/CRT-Ds: pre-defined device programming, measurements and follow-up schedule
  Plexa S DX: Implantation, measurements and follow-up schedule
Period: Overall Study
Arm/Group | Acticor/Rivacor ICDs/CRT-Ds
Started | 130
Patients With Implantation Attempt | 128
Patients Implanted | 127
Completed | 111
Not Completed | 19
Not completed — Death | 5
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 4
Not completed — Device explanted | 3
Not completed — No study device implanted | 3

BASELINE CHARACTERISTICS:
Population: Of 130 enrolled patients, 128 underwent an implantation attempt with an investigational device (COR family ICD or Plexa S DC lead) and were included in the baseline analysis population. Two patient received a non-investigational device and were therefore excluded in the baseline analysis.
Arm/Group | Acticor/Rivacor ICDs/CRT-Ds
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 102
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 13
  Latvia | 17
  Netherlands | 21
  Hungary | 24
  Slovakia | 4
  Switzerland | 22
  Germany | 27

OUTCOME MEASURES:

1. Primary Outcome: Cor Family-related Serious Adverse Device Effect (SADE)-Free Rate Until 3-month Follow-up
Description: Serious Adverse Device Effect (SADE)-free rate possibly or securely related to the Cor Family Internal Cardioverter Defibrillators (ICDs) / Cardiac Resynchronisation Therapy-Defibrillators (CRT-Ds) until 3-month follow-up
Time Frame: 3 months
Population: All patients who either had a primary endpoint or who had reached 3 months of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Acticor/Rivacor ICDs/CRT-Ds
Number analyzed (Participants) | 123
Participants | 122
Statistical Analysis 1: Comparison: Acticor/Rivacor ICDs/CRT-Ds; Serious Adverse Device Effects (SADE) possibly or securely related to the Cor Family devices until the 3- month follow-up are counted for this primary endpoint. The following hypothesis has been defined: Ho: SADE-free rate through 3 months post-implant ≤ 90.0% Ha: SADE-free rate through 3 months post-implant > 90.0%; Test type: Other — No comparison of two groups, just single arm design; p = 0.05, t-test, 2 sided; SADE-free rate in the study group = 0.98, 95% CI 2-sided [0.9 to 1]

2. Secondary Outcome: Kaplan-Meier Estimate for the Cor Family Related SADE-free Rate
Description: Application of the Kaplan-Meier method to estimate the 3-month (92 days) SADE-free rate and the 12-month (365 days) SADE-free rate
Time Frame: 3 months, 12 months
Population: Of 130 enrolled patients, 127 implanted with a COR Family ICD. Out of these, 123 patients were eligible for these endpoint analysis; 4 patients had premature study termination before day 61 after implantation without experiencing a Serious Adverse Device Effect related to the Cor Family device (SADE-d) and were excluded from analysis. For the 12-month endpoint, 111 patients who completed the study were eligible for endpoint analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Kaplan-Meier-Estimate for the Cor-Family Related SADE-free Rate 92 Days After Implantation: Implant of the new Cor Family ICDs and Plexa ProMRI S DX lead (if applicable). Device measurements, pre-defined programming and Adverse Event Reporting
  Acticor/Rivacor ICDs/CRT-Ds: pre-defined device programming, measurements and follow-up schedule
  Plexa S DX: Implantation, measurements and follow-up schedule
- Kaplan-Meier-Estimate for the Cor-Family Related SADE-free Rate 365 Days After Implantation: Implant of the new Cor Family ICDs and Plexa ProMRI S DX lead (if applicable). Device measurements, pre-defined programming and Adverse Event Reporting.
  Acticor/Rivacor ICDs/CRT-Ds: pre-defined device programming, measurements and follow-up schedule
  Plexa S DX: Implantation, measurements and follow-up schedule
Arm/Group | Kaplan-Meier-Estimate for the Cor-Family Related SADE-free Rate 92 Days After Implantation | Kaplan-Meier-Estimate for the Cor-Family Related SADE-free Rate 365 Days After Implantation
Number analyzed (Participants) | 123 | 111
percentage of participants | 99.2 [94.5 to 99.9] | 99.2 [94.5 to 99.9]
Statistical Analysis 1: Comparison: Kaplan-Meier-Estimate for the Cor-Family Related SADE-free Rate 92 Days After Implantation vs Kaplan-Meier-Estimate for the Cor-Family Related SADE-free Rate 365 Days After Implantation; Test type: Other — Kaplan-Meier method; The Kaplan-Meier method will be applied to estimate the 3-month SADE-free rate at 92 days after implantation (sensitivity analysis of the primary endpoint) and the 12-month SADE-free rate at 365 days after implantation

3. Secondary Outcome: Number of Handling-Assessments of the Automatic LV VectorOpt Test (CRT-devices Only) by the Investigator
Description: Investigators were asked to assess the overall handling of the Automatic LV VectorOpt test in patients who received a CRT-device. Assessments were collected during implantation, pre-hospital discharge, and 3-month follow-up visit. The following options could be chosen by the investigator: Very good - good - adequate - poor -very poor.
Time Frame: 3 months
Population: In total, 52 assessments were received from the investigators: 24 assessments at time of implantation, 21 assessments at time of pre-hospital discharge, 7 assessments during 3-month follow-up visit
Measure: Number; unit: Handling-assessment by investigator
Units Other Than Participants: handling-assessments
Arm/Group | Acticor/Rivacor ICDs/CRT-Ds
Number analyzed (Participants) | 52
Number analyzed (handling-assessments) | 52
Handling-assessment by investigator
  Very good | 21
  Good | 27
  Adequate | 3
  Poor | 1
  Very poor | 0

4. Secondary Outcome: Number of Handling-Assessments for the Overall Handling of the CRT AutoAdapt Feature (CRT-devices Only) by the Investigator
Description: Investigator were asked to assess the overall handling of the CRT AutoAdapt feature in patients who received a CRT-device. Assessments were collected during the 3-month follow-up visit.
  The following options could be chosen by the investigator: Very good - good - adequate -poor -very poor.
Time Frame: 3 months
Population: In total, 20 assessments were received from the investigator at the time of the 3-month follow-up visit.
Measure: Number; unit: Handling-assessment by investigator
Units Other Than Participants: handling-assessments
Arm/Group | Acticor/Rivacor ICDs/CRT-Ds
Number analyzed (Participants) | 20
Number analyzed (handling-assessments) | 20
Handling-assessment by investigator
  Very good | 7
  Good | 10
  Adequate | 3
  Poor | 0
  Very poor | 0

ADVERSE EVENTS:
Time Frame: Patients were followed for 1 year
Arm/Group | Acticor/Rivacor ICDs/CRT-Ds
All-Cause Mortality (participants affected / at risk) | 5/130
Serious Adverse Events (participants affected / at risk) | 54/130
Other Adverse Events (participants affected / at risk) | 42/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acticor/Rivacor ICDs/CRT-Ds (N=130)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Adverse drug reaction (General disorders) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Aortic intramural haematoma (Vascular disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 9 (13)
Cardiac failure chronic (Cardiac disorders) | 2 (2)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Crepitations (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Device connection issue (Product Issues) | 1 (1)
Device electrical impedance issue (Product Issues) | 1 (1)
Device lead damage (Product Issues) | 1 (1)
Device pacing issue (Product Issues) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastric dysplasia (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (3)
Hypothyroidism (Endocrine disorders) | 1 (1)
Implant site haematoma (General disorders) | 2 (2)
Implant site haemorrhage (General disorders) | 1 (1)
Implantation complication (Injury, poisoning and procedural complications) | 1 (1)
Inflammation (General disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1)
Lead dislodgement (Product Issues) | 1 (1)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 3 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Postoperative hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 2 (2)
Psychomotor skills impaired (Nervous system disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 2 (2)
Renal disorder (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Sensing amplitude decreased (Product Issues) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ventricular dyssynchrony (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 4 (7)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acticor/Rivacor ICDs/CRT-Ds (N=130)
Adverse drug reaction (General disorders) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Cardiac vein dissection (Injury, poisoning and procedural complications) | 1 (1)
Chest pain (General disorders) | 2 (2)
Circulatory collapse (Vascular disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Complication of device insertion (General disorders) | 1 (1)
Condition aggravated (General disorders) | 2 (2)
Corona virus infection (Infections and infestations) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Device computer issue (Product Issues) | 1 (1)
Device inappropriate shock delivery (Product Issues) | 1 (1)
Device stimulation issue (Product Issues) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)
Electromagnetic interference (Product Issues) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Implant site haematoma (General disorders) | 4 (4)
Implant site inflammation (General disorders) | 1 (1)
Implant site pain (General disorders) | 2 (2)
Implant site swelling (General disorders) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Oversensing (Product Issues) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Undersensing (Product Issues) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT03891329/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03891329/SAP_001.pdf